CLINICAL TRIAL: NCT03748797
Title: Effects of Supervised Exercise Program on Physical Health and Quality of Life Among Older Adults Living With HIV in Hong Kong
Brief Title: Effects of Supervised Exercise on Physical Health and Quality of Life Among Older HIV Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Society for AIDS Care (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hong, CHUNG, Physiotherapist, The Society for AIDS Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: supervised exercise
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: HIV/AIDS
Keywords: HIV, exercise, aging, physical health, quality of life
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Exercise group: Performed an 8-week, 2 times/week exercise training (moderate intensity) under physiotherapist supervision.
  Control group: No supervised exercise training given. Participants were advised to continue their routine daily activities and self exercises if they have.
Who Masked: Outcomes Assessor
Masking Description: A research assistant who was blinded for the participants grouping was responsible for data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): 8-week moderate intensity exercise training under supervision
  Interventions: Other: Moderate intensity exercise training under supervision
- Control group (No Intervention): No supervised exercise training given. Participants were advised to continue their routine daily activities and self exercises if they have

INTERVENTIONS:
Other: Moderate intensity exercise training under supervision — Upper and lower limbs cycling, treadmill walking, multi-gym strengthening, stepper exercise, dumb bell and squatting exercise
  Arms: Exercise group

SUMMARY:
The effects of exercise for older HIV-infected adults have not been well studied, especially in Chinese population. This study aimed to investigate the effect of supervised exercise on physical health and quality of life among older people living with HIV (PLWH) in Hong Kong.

HIV-infected adults were recruited from a community-based Non-Governmental Organization (NGO) for HIV patient services. Participants were randomized into exercise group or control group. The participants in exercise group performed an 8-week moderate intensity supervised exercise program. In the control group, participants were not given any supervised exercises. They were advised to continue their routine daily activities and self exercises.

Outcomes were measured for both groups at baseline and after 8 weeks. Primary outcomes: grip strength, 30 seconds chair stand, 6 minutes-walk test and Short Form-36 questionnaire (SF-36). Secondary outcome: Subjective improvement

At the end of the program, all participants from exercise group were interviewed individually by principle investigator to allow feedbacks.

DETAILED DESCRIPTION:
It is a randomized controlled trial. HIV-infected adults were recruited from a community-based Non-Governmental Organization (NGO) for HIV patient services.They were randomized into exercise group or control group by drawing lots which contained equal number of orange balls (exercise) and white balls (control)

The participants in exercise group performed an 8-week, 2 times/week supervised exercise program in the community day center of the recruiting NGO. Exercise sessions were organized in a group of 2 to 3 participants. The exercises were supervised by a registered physiotherapist to ensure exercise safety and quality. Exercise intensity was moderate. We monitored the heart rate of participants during exercise and maintained around 50% to 70% of maximum heart rate. Blood pressure and oxygen saturation were also checked for safety purposes. The mode of exercise was combined aerobic and resistance training. It involved upper and lower limbs cycling, treadmill walking, multi-gym strengthening, stepper exercise, dumb bell and squatting exercise. The duration for each exercise session was around 45 minutes. Duration and intensity of exercises were adjusted depending on the tolerance and physical capacity of each participant. In the control group, participants were not given any supervised exercises. They were advised to continue their routine daily activities and self exercises. Control group participants were allowed to join into the same training program after the research had finished.

Outcomes were measured for both groups at baseline and after 8 weeks in the same community day center. A research assistant who was blinded for the participants grouping was responsible for data collection. Physical health parameters included grip strength, 30 seconds chair stand and 6 minutes-walk test. Health related quality of life was measured by Short Form-36 questionnaire (SF-36). Subjective improvement was taken in form of Likert scale, from -100% to +100% with 10% interval in each possible response.

At the end of the program, all participants from exercise group were interviewed individually by principle investigator to allow feedbacks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with HIV age > 50, treating with antiretroviral therapy
2. No contraindication to moderate intensity exercise
3. Independent Outdoor walker without assistance
4. Sedentry participants who have not received any structural / supervised exercise program in the past 1 year

Exclusion Criteria:

1. Age <50
2. Unstable or unfit for exercise
3. Wheelchair user or assisted walker
4. Already had regular exercise habit or under structural exercise program in the past 1 year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change of SF-36 scores | Change from Baseline SF-36 scores at 8 weeks
  Short Form 36 (SF-36) questionnaire is used to assess health related quality of life
Change of Grip strength | Change from Baseline grip strength at 8 weeks
  Maximum grip strength of the participant in kg
Change of 30 seconds chair stand | Change from Baseline performance at 8 weeks
  Number of times that the participant stand up and sit down within 30 seconds
Change of 6 minutes walk test | Change from Baseline performance at 8 weeks
  The distance (in meters) which the participant is able to walk in 6 minutes

SECONDARY OUTCOMES:
Subjective improvement | Subjective change after 8 weeks compare to baseline
  Subjective physical improvement reported by participant (from -100% to +100%)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hong Chung, MSc, Principal Investigator — The Society for AIDS Care
Locations (1):
- The Society for AIDS Care Day Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided